CLINICAL TRIAL: NCT01502033
Title: An Open-Label Eight-Week Trial of Repetitive Transcranial Magnetic Stimulation in Depressed Adolescents: Mechanisms of Response
Brief Title: Study of Repetitive Transcranial Magnetic Stimulation (rTMS) in Depressed Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paul E. Croarkin (Other)
Responsible Party: Sponsor-Investigator, Paul E. Croarkin, Assistant Professor of Child and Adolescent Psychiatry, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-004500
Record Dates: First submitted 2011-12-27; First posted 2011-12-30 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Major Depressive Disorder
Keywords: Adolescent Depression; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transcranial Magnetic Stimulation (Experimental): Open-label course of 30 daily treatments with repetitive transcranial magnetic stimulation (rTMS) at 120% magnetic field intensity relative to the patient's resting motor threshold, at 10 pulses per second (10 Hz) for 4 seconds, with an intertrain interval of 26 seconds for a total of 75 trains per treatment session.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — 30 daily treatments of (over 6-8 weeks) of 10 Hz rTMS at 120% motor threshold, applied to the left dorsolateral prefrontal cortex with 3,000 stimulations per treatment
  Other Names: NeuroStar

SUMMARY:
This research study aims to test the safety and effectiveness of repetitive transcranial magnetic stimulation (rTMS) on teens with depression. The study also seeks to understand how rTMS treatment affects the neurobiology of teens with depression.

DETAILED DESCRIPTION:
This study aims to:

1. Evaluate the antidepressant effect and safety of rTMS in adolescents meeting criteria for major depressive disorder, single or recurrent episode.
2. Evaluate, by proton magnetic resonance spectroscopy (1H-MRS) at 3 Tesla (3T), the regional specificity [anterior cingulate (AC) vs. left dorsolateral prefrontal cortex (L-DLPFC)] of cerebral metabolites (glutamate and glutamine) in adolescent depression and study whether glutamine resonances are associated with response or remission of clinical depressive symptoms when rTMS is used to treat adolescent depression.
3. Evaluate the accuracy of an efficient method for locating the F3 position (i.e., L-DLPFC) through comparison with magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unipolar major depressive disorder, in a current major depressive episode, without psychotic features
* Pretreatment CDRS-R Raw score ≥ 40
* Age is at least 13 and less than 19 years
* Ongoing, stable dose antidepressant therapy for at least 6 weeks to include the following antidepressants (with dosing range):

  * Celexa (citalopram hydrobromide) - 10 to 60mg
  * Cymbalta (duloxetine) - 40mg to 120mg
  * Desyrel (trazodone HCl) - 12.5mg to 150mg
  * Effexor (venlafaxine HCl) - 37.5mg to 300mg
  * Luvox (fluvoxamine maleate) - 25mg to 200mg
  * Lexapro (escitalopram oxalate) - 10mg to 40mg
  * Paxil (paroxetine HCl) - 10mg to 50mg
  * Pristiq (desvenlafaxine) - 50mg to 100mg
  * Prozac (fluoxetine HCl) - 10mg to 80mg
  * Remeron (mirtazapine) - 7.5mg to 45mg
  * Zoloft (sertraline HCl) - 25mg to 200mg
* Subjects able to attend at least 31 study visits at Mayo Clinic - Rochester
* Willing to provide informed assent (adolescent) and informed consent (family)

Exclusion Criteria:

* Subjects currently on stimulant, antipsychotic, bupropion or tricyclic antidepressant medications.
* Prior rTMS, vagus nerve stimulation (VNS) or electroconvulsive therapy (ECT)
* Contraindication to MRI
* Contraindication to rTMS (history of neurological disorder such as seizures, increased intracranial pressure, brain surgery, or head trauma with loss of consciousness for >15 minutes, history of stroke, family history of epilepsy, intracardiac lines, Anticoagulant, immune suppressive and/or chemotherapy, or those who received any of these therapies within 3 months before enrollment in the study Unstable medication conditions such as hematological or infectious (e.g., human immunodeficiency virus-HIV) disorders, implanted electronic device, metal in the head, or pregnancy)
* History of schizophrenia, schizoaffective disorder, other [non mood disorder] psychosis, depression secondary to a medical condition, mental retardation, substance dependence or abuse within the past year (except nicotine), bipolar disorder, psychotic features in this or previous episodes, amnestic disorder, obsessive compulsive disorder, post-traumatic stress disorder, panic disorder
* History of autoimmune, endocrine, viral, or vascular disorder.
* Unstable cardiac disease, uncontrolled hypertension, or sleep apnea
* Active suicidal intent or plan, or history of attempt within the past 6 months

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Croarkin, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wall CA, Croarkin PE, McClintock SM, Murphy LL, Bandel LA, Sim LA, Sampson SM. Neurocognitive effects of repetitive transcranial magnetic stimulation in adolescents with major depressive disorder. Front Psychiatry. 2013 Dec 12;4:165. doi: 10.3389/fpsyt.2013.00165. eCollection 2013. PMID 24376426
- [Derived] Sonmez AI, Kucuker MU, Lewis CP, Kolla BP, Doruk Camsari D, Vande Voort JL, Schak KM, Kung S, Croarkin PE. Improvement in hypersomnia with high frequency repetitive transcranial magnetic stimulation in depressed adolescents: Preliminary evidence from an open-label study. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Mar 8;97:109763. doi: 10.1016/j.pnpbp.2019.109763. Epub 2019 Oct 18. PMID 31634515
- [Derived] Wall CA, Croarkin PE, Maroney-Smith MJ, Haugen LM, Baruth JM, Frye MA, Sampson SM, Port JD. Magnetic Resonance Imaging-Guided, Open-Label, High-Frequency Repetitive Transcranial Magnetic Stimulation for Adolescents with Major Depressive Disorder. J Child Adolesc Psychopharmacol. 2016 Sep;26(7):582-9. doi: 10.1089/cap.2015.0217. Epub 2016 Feb 5. PMID 26849202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 participants recruited(and enrolled) from the Mayo Clinic Child and Adolescent Mood Disorders Clinic.
Pre-assignment Details: Participants were maintained on stable dosage of antidepressant medication for 4 weeks prior to enrollment and rTMS treatment.
Groups:
- Transcranial Magnetic Stimulation: Open-label course of 30 daily treatments with repetitive transcranial magnetic stimulation (rTMS) at 120% magnetic field intensity relative to the patient's resting motor threshold, at 10 pulses per second (10 Hz) for 4 seconds, with an intertrain interval of 26 seconds for a total of 75 trains per treatment session.
  Transcranial Magnetic Stimulation
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation
Started | 10 (Milestone (10 participants) met.)
Completed | 7 (Milestone (10 participants) met)
Not Completed | 3
Not completed — 1 participant had scalp discomfort | 1
Not completed — 1 participant had worsening depression | 1
Not completed — 1 participant went back to school | 1

BASELINE CHARACTERISTICS:
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.9 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10
Children's Depression Rating Scale Revised [Median (Standard Deviation); unit: units on a scale] — Range of total score is 17-113 Total score of 40 or higher indicates moderate to severe depression (higher scores indicate increased severity of depressive symptoms).
  A score below 40 indicates mild or minimal depressive symptoms.
  units on a scale | 62.9 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Children's Depression Rating Scale-Revised (CDRS-R) Post Treatment 30 or Last Treatment (in Cases of Early Withdrawal)
Description: The Children's Depression Rating Scale-Revised (CDRS-R) is a validated, 17-item, semi-structured clinician rating tool to assess severity of depression with subject and parental input for 14 of the 17 items.
Time Frame: 5 days of Treatment 30 or Last Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10
units on a scale | 41.8 (13.2)

2. Secondary Outcome: Clinical Global Impression - Severity (CGI-S) Post Treatment 30 or Last Treatment (in Cases of Early Withdrawal)
Description: The Clinical Global Impression - Severity (CGI-S) is a standardized assessment utilizing a 7-point scale with which the clinician rates severity of the subject's depressive illness at the time of assessment relative to the clinician's past experience with patients with the same diagnosis. Range of scale is 1-7 (1= normal, not ill at all; 7= among the most ill patients; larger number indicates greater severity of symptoms or worse outcome).
Time Frame: Within 5 days of Treatment 30 or Last Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open Label Active Treatment: All participants had unblended treatment
Arm/Group | Open Label Active Treatment
Number analyzed (Participants) | 10
units on a scale | 3.4 (1.5)

3. Secondary Outcome: The Clinical Global Impression - Improvement (CGI-I)
Description: The Clinical Global Impression - Improvement (CGI-I) is a standardized assessment utilizing a 7-point scale with which the clinician rates improvment of the subject's depressive illness at the time of assessment relative to the clinician's past experience with patients with the same diagnosis. Range of scale is 1-7 (1= very much improved, 7=very much worse) larger number indicates greater severity of symptoms or worse outcome).
Time Frame: Within 5 days of 30 treatments or after last treatment in case of early withdrawal
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Magnetic Stimulation
Number analyzed (Participants) | 10
units on a scale | 2.7 (1.1)

ADVERSE EVENTS:
Groups:
- Open Label Active Treatment: All participants had unblinded treatment
Arm/Group | Open Label Active Treatment
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Active Treatment (N=10)
scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) — One participant had scalp pain with the initial session and discontinued treatment.
Anxiety (Psychiatric disorders) | 1 (1) — Anxiety (related to school expectations)
Depression (Psychiatric disorders) | 1 (1) — Worsening depression

LIMITATIONS AND CAVEATS:
Please note that clinical results must be interpreted with caution due to small sample size and study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No